CLINICAL TRIAL: NCT01490541
Title: The Predictive Scores for Gastric Cancer in Gastric Intestinal Metaplasia (GIM) Patient: a Recommendation for Thai Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Principle investigator, King Chulalongkorn Memorial Hospital
Other Study IDs: RP003
Record Dates: First submitted 2011-12-05; First posted 2011-12-13 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Gastric Intestinal Metaplasia
Keywords: Gastric intestinal metaplasia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gastric intestinal metaplasia patient

SUMMARY:
The predictive scores for gastric cancer in gastric intestinal metaplasia(GIM) patient: a recommendation for Thai population.

Objective:

To evaluate major risk factors for gastric cancer in gastric intestinal metaplasia(GIM) patient in order to propose the appropriate recommendation for Thai people.

Research Design:

Single center, retrospective-cohort study.

DETAILED DESCRIPTION:
Study population and Sample size at Faculty of Medicine, Chulalongkorn University The patients who were diagnosed gastric intestinal metaplasia from 1997 to 2012 and then follow up for 5 years. Estimate sample size =280

* Investigational product, dosage & route of administration
* Questionnaire for explore the risk factors
* EGD with biopsy
* Blood sampling for gastro panel
* Duration of participation
* 5 years or until diagnose gastric cancer

Statistical method:

Unconditional-binary-logistic regression

ELIGIBILITY:
Inclusion Criteria:

1. All patients were diagnosed GIM
2. All patients have to sign the consent form

Exclusion Criteria:

1. Previous gastric surgery including gastrectomy and bypass surgery
2. Bleeding tendency including decompensated cirrhosis, chronic kidney disease and long-tem antiplatelets or anticoagulants
3. HIV infection
4. History of proton pump inhibitor use within 1 week
5. History of antibiotic use within 4 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All GIM patients in KCMH whose diagnosed from 1997 to 2005, at least 280.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The prevalence of early gastric cancer in gastric intestinal metaplasia(GIM) patient from 5 year-follow-up in Thai population | Up to 5 years
  In Thailand, gastric cancer patients usually presented with advance stage and carried the dismal prognosis. GIM is a well known precancerous lesion. The appropriate follow-up period in high risk GIM patient can increase the prevalence of early gastric cancer and reduce the mortality rate of gastric cancer

CONTACTS AND LOCATIONS:
Overall Officials: Rungsun Rerknimitr, Professor, Study Director — King Chulalongkorn Memorial Hospital; Rapat Pittayanon, MD, Principal Investigator — King Chulalongkron Memorial Hospital
Locations (1):
- Rapat Pittayanon, Bangkok, Bangkok, Thailand

REFERENCES:
- See also: Ethic committee of KCMH — http://www.medchulairb.com